CLINICAL TRIAL: NCT00399711
Title: Repaglinide and Metformin Combination Tablet (NN4440) in a TID Regimen Compared to a BID Regimen and BID Avandamet in Subjects With Type 2 Diabetes: A Twenty-Six Week, Open-Label, Multicenter, Randomized, Parallel Group Trial to Investigate Efficacy and Safety
Brief Title: Effect of Repaglinide and Metformin Combination Tablet or Rosiglitazone and Metformin in Fixed Dose Combination on Blood Glucose Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN4440-1794
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: repaglinide and metformin combination tablet
Drug: rosiglitazone and metformin combination tablet

SUMMARY:
This trial is conducted in the United States of America (USA). This trial compares the changes in HbA1c after 26 weeks of repaglinide and metformin fixed dose combination tablet given as twice daily versus three times daily regimens or versus twice daily rosiglitazone and metformin fixed dose combination tablet in subjects with type 2 diabetes currently on monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 3 months
* HbA1c between 7.5-11.0% on monotherapy or
* HbA1c between 7.0-10.0% on dual therapy
* BMI maximum 45 kg/m2

Exclusion Criteria:

* Any clinically significant disease history in the opinion of the investigator
* Severe heart disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 26 weeks of treatment

SECONDARY OUTCOMES:
Change in 8-point Glucose Profiles
Change in Lipid Profile
Events of hypoglycemia
Safety parameters
Change in Fasting Plasma Glucose
Waist/hip ratio change
Change in body weight
Percentage of subjects achieving sudden levels of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), MD, Study Director — Novo Nordisk A/S
Locations (94):
- United States (93):
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Jonesboro, Arkansas
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Redlands, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Hamden, Connecticut
  - Novo Nordisk Investigational Site, Stamford, Connecticut
  - Novo Nordisk Investigational Site, Aventura, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Daytona Beach, Florida
  - Novo Nordisk Investigational Site, Inverness, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Longwood, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Aurora, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Flossmoor, Illinois
  - Novo Nordisk Investigational Site, Naperville, Illinois
  - Novo Nordisk Investigational Site, Oak Brook, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Vernon Hills, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Des Moines, Iowa
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Erlanger, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Bossier City, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Oak Park, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Jersey City, New Jersey
  - Novo Nordisk Investigational Site, Warren Township, New Jersey
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Springfield, Pennsylvania
  - Novo Nordisk Investigational Site, Cranston, Rhode Island
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Henrico, Virginia
  - Novo Nordisk Investigational Site, Lebanon, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Novo Nordisk Investigational Site, San Juan, Puerto Rico

REFERENCES:
- [Result] Raskin P, Lewin A, Reinhardt R, Lyness W; Repaglinide/Metformin Fixed-Dose Combination Study Group. Twice-daily and three-times-daily dosing of a repaglinide/metformin fixed-dose combination tablet provide similar glycaemic control. Diabetes Obes Metab. 2009 Oct;11(10):947-52. doi: 10.1111/j.1463-1326.2009.01069.x. Epub 2009 Jun 16. PMID 19531054
- [Result] Raskin P, Lewin A, Reinhardt R, Lyness W; Repaglinide/Metformin Fixed-Dose Combination Study Group. Twice-daily dosing of a repaglinide/metformin fixed-dose combination tablet provides glycaemic control comparable to rosiglitazone/metformin tablet. Diabetes Obes Metab. 2009 Sep;11(9):865-73. doi: 10.1111/j.1463-1326.2009.01062.x. Epub 2009 May 19. PMID 19476470
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com